CLINICAL TRIAL: NCT02031250
Title: Randomized Phase II Study of DCE-MRI-based Dose Escalation for Poor-prognosis and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.062; HUM00074305 (Other: University of Michigan)
Record Dates: First submitted 2013-12-12; First posted 2014-01-09 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Active Comparator): Standard chemotherapy (Cisplatin or Carboplatin) and IMRT (Intensity-Modulated Radiation Therapy)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Radiation: IMRT (Intensity-Modulated Radiation Therapy)
- Boost Arm (Experimental): Boost radiation to hypoperfused/low-diffusion volumes in addition to standard chemotherapy (Cisplatin or Carboplatin) and IMRT (Intensity-Modulated Radiation Therapy)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Radiation: IMRT (Intensity-Modulated Radiation Therapy); Radiation: Boost Radiation to Hypoperfused Volumes

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 40mg/m2 administered as an IV infusion prior to radiotherapy on day 1 of each week of chemo-irradiation
Drug: Carboplatin — Patients considered medically unfit to receive Cisplatin as determined by the prescribing physician, will receive Carboplatin via IV infusion on day 1 of each week of chemo-irradiation
Radiation: IMRT (Intensity-Modulated Radiation Therapy)
Radiation: Boost Radiation to Hypoperfused Volumes
  Arms: Boost Arm

SUMMARY:
This study aims to improve locoregional control of poor prognosis Head and Neck Cancer (HNC) patients by selectively escalating the radiotherapy dose to subvolumes of tumor likely to be resistant to standard Radiation Therapy (RT) using DCE-MRI (Dynamic Contrast Enhanced Magnetic Resonance Imaging). Standard doses of radiotherapy to the rest of the tissues and surrounding normal tissues will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, non-metastatic locally/regionally advanced squamous cell carcinoma of the head and neck, stage III/IV, referred for definitive chemo-RT, and meet one of the following six criteria:

  1. Primary tumor (T4) with or without metastatic lymph nodes. Tumor or nodes are: unresectable, resection is considered by the treating surgeon or patient to result in unacceptable functional or oncological results, patient refuses surgery, or surgery is not possible due to comorbidities.
  2. HPV(-) (Human Papillomavirus) or p16(-) locally/regionally advanced (T3-4 or N2-3) oropharyngeal cancer.
  3. HPV(+) or p16(+) locally/regionally advanced (T4 or N3) oropharyngeal cancer.
  4. T3 or T4 laryngeal or hypopharyngeal cancer that is locally advanced, bulky (>40 cc*), unresectable, or patient declines surgery.
  5. Stage III/IV oral cavity or paranasal sinus cancers in patients who refuse surgery or are unfit for surgery.
  6. Locally/regionally advanced (stage T3-4 and/or N3) nasopharyngeal cancer which is EBV (-) (Epstein-Barr Virus).
* KPS (Karnofsky Performance Status: A measure of general well being and activities of daily living; scores range from 0 to 100 where 100 represents perfect health) >70 (see Appendix A) within two weeks of enrollment.
* Pre-treatment laboratory criteria within four weeks of enrollment:

  * WBC (White Blood Cell) > 3500/ul, granulocyte > 1500/ul.
  * Platelet count > 100,000/ul.
  * Total Bilirubin < 1.5 X ULN.
  * AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) < 2.5 X ULN.
  * Estimated Creatinine clearance >30cc/min.
* Patients must be able to receive protocol chemotherapy in the judgment of the treating Medical Oncologist.
* Patients are adults (Age ≥18).
* All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* EBV (+) Nasopharyngeal Carcinoma in the protocol treated tumor.
* Prior head and neck radiation.
* Documented evidence of distant metastases.
* Patients with active infection.
* Pregnant women.
* Patients should have no contraindications to having a contrast enhanced MRI scan. These contraindications will be assessed at the time of enrollment using the guidelines set up and in clinical use by the Institutional Standard Practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DSF) time | 3 years post treatment
  Kaplan-Meier curves with point-wise 90% confidence intervals will be generated for each treatment arm, overall and by strata. Estimates with confidence intervals will be generated from these curves for the usual summary statistics, including median DFS times and DFS at 1, 2, and 3 years.

SECONDARY OUTCOMES:
Local-regional control rate | 3 years post-treatment
  Compare local-regional control rates between the two arms at 1, 2 and 3 years. Local-regional control is defined as the absence of local-regional progression.
Proportion of patients in which hypoperfused/low-diffusion subvolumes overlap with recurrence volumes | 3 years post treatment
Number of patients with adverse events | 3 years post treatment
  Acute and late toxicities will be summarized descriptively by grade and type for each treatment group. The proportion of patients experiencing certain toxicity types will be calculated with score based confidence intervals. Chi-square tests will be used to test whether the proportion of patients with toxicity differs between treatment groups.
Correlation coefficient between continuous dose and perfusion summary measures | 2 weeks post Radiation Therapy (RT)
  Pearson or Spearman rank based correlation between the continuous dose and perfusion summary measures

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - Veterans Affairs (VA) Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Hospital, Ann Arbor, Michigan